CLINICAL TRIAL: NCT04087031
Title: Assistive Robotic in the Elderly: Innovative Models in the Rehabilitation of the Elderly With Parkinson's Disease Through Technological Innovation
Brief Title: Innovative Models in the Rehabilitation of the Elderly With Parkinson's Disease Through Technological Innovation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INRCA_02_2019
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease; Frail Elderly; Robotic Devices in Rehabilitation
Keywords: Parkinson disease; robotics; elderly; rehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control arm (Active Comparator): Ten traditional treatment sessions divided into 2 training sessions per week for 5 weeks
  Interventions: Other: control arm
- virtual reality games arm (Experimental): Ten technological treatment sessions divided into 2 training sessions per week for 5 weeks
  Interventions: Other: virtual reality games
- robotic treadmill arm (Experimental): Ten technological treatment sessions divided into 2 training sessions per week for 5 weeks
  Interventions: Other: robotic treadmill

INTERVENTIONS:
Other: control arm — Each session will include 50 minutes of traditional physical rehabilitation therapy
  Arms: control arm
Other: virtual reality games — Each session will include 30 minutes of traditional physical rehabilitation therapy followed by 20 minutes of robotic Tymo system (Tyromotion, Austria), a wireless static and dynamic platform, for evaluating and rehabilitating posture.
  Arms: virtual reality games arm
Other: robotic treadmill — Each session will include 30 minutes of traditional physical rehabilitation therapy followed by 20 minutes of robotic Walker View (TecnoBody, Italy) a treadmill equipped with a sensorized belt with eight load cells and a 3D camera
  Arms: robotic treadmill arm

SUMMARY:
The final goal of the present study is to propose a new approach in the Parkinson's Disease rehabilitation, focused on the use of robotic devices and to check the results not only at the end of the treatment but also in the long term, foreseeing 3 follow-up.

DETAILED DESCRIPTION:
Parkinson's disease is one of the most frequent causes of disability among the elderly. It is a chronic-progressive neuro-degenerative disease, characterized by several motor disorders. The balance disorder is a symptom that involves the body axis; it is due to a reduction in the straightening reflexes, so the subject is not able to correct any imbalances. Balance disorders do not respond to dopaminergic therapy used in Parkinson's disease. Therefore, physiotherapy becomes an important intervention for the management of motor disorders. Originally, these rehabilitative approaches were based on empirical experiences, but several scientific evidence suggests that neuronal plasticity is exercise-dependent. In this context, robotic rehabilitation performs an important role because it allows to perform task-oriented exercises and to increase the number of repetitions and their intensity. This protocol study aims to evaluate an innovative rehabilitation treatment of the elderly patients with Parkinson's disease, designed to improve the gait and to reduce the risk of falling. The treatment involves the use of two robotic devices: Tymo system and Walker View.

This study is a single-blinded randomized controlled trial. 195 patients with PD will be recruited and randomly divided into three groups, to receive a traditional rehabilitation program or a robotic rehabilitation using Tyro system or Walker View in addition to the traditional therapy. Assessments will be performed at baseline, at the end of treatment and 6 months, 1 year and 2 years from the end of the treatment. A 10 treatment sessions will be conducted, divided into 2 training sessions per week, for 5 weeks. The control group will perform traditional therapy sessions lasting 50 minutes. The technological intervention group will carry out 30 minutes of traditional therapy and 20 minutes of treatment with a robotic system.

ELIGIBILITY:
Inclusion Criteria:

* Hoen and Yahr scale: 1-3 stage
* FAC ≤ 2
* Ranking scale score ≤ 3
* Stability of drug treatment for at least 1 month
* Geriatric Depression Scale 5-items: negative

Exclusion Criteria:

* Concomitant participation in other studies
* Lack of written informed consent
* Clinical dementia rating (CDR) score ≥ 3
* History of syncopal episodes, epilepsy and vertigo not controlled pharmacologically
* Serious dysfunction of the autonomic system
* Severe behavioral syndromes not compensated by drugs
* Concurrent neurological diseases
* Severe systemic diseases with life expectancy < 1 year
* Patients unable to follow up.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2019-12-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
difference in falling risk among virtual reality games arm, robotic treadmill arm and control arm | before treatment, at the end of treatment and 6, 12 and 24 months after the end of treatment
  falling risk will be evaluated by the Tinetti performance oriented mobility assessment (POMA). POMA test has two subscales, Balance and Gait sections. Total score is obtained by adding the scores of the two subscales (balance + gait) . Total score < 19 high fall risk, total score 19-24 medium fall risk, total score 25-28 low fall risk.

SECONDARY OUTCOMES:
difference in gait performance among virtual reality games arm, robotic treadmill arm and control arm | before treatment, at the end of treatment and 6, 12 and 24 months after the end of treatment
  gait performance will be assessed by walking speed through instrumental Gait Analysis
difference in fear of falling among virtual reality games arm, robotic treadmill arm and control arm | before treatment, at the end of treatment and 6, 12 and 24 months after the end of treatment
  fear of falling will be evaluated by the Falls Efficacy Scale - International (FES-I). Higher scores represent greater the fear of falling (ranging from 16 to 64)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS INRCA Hospital, Ancona
  - IRCCS INRCA Hospital, Fermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maranesi E, Casoni E, Baldoni R, Barboni I, Rinaldi N, Tramontana B, Amabili G, Benadduci M, Barbarossa F, Luzi R, Di Donna V, Scendoni P, Pelliccioni G, Lattanzio F, Riccardi GR, Bevilacqua R. The Effect of Non-Immersive Virtual Reality Exergames versus Traditional Physiotherapy in Parkinson's Disease Older Patients: Preliminary Results from a Randomized-Controlled Trial. Int J Environ Res Public Health. 2022 Nov 10;19(22):14818. doi: 10.3390/ijerph192214818. PMID 36429537
- [Derived] Bevilacqua R, Maranesi E, Di Rosa M, Luzi R, Casoni E, Rinaldi N, Baldoni R, Lattanzio F, Di Donna V, Pelliccioni G, Riccardi GR. Rehabilitation of older people with Parkinson's disease: an innovative protocol for RCT study to evaluate the potential of robotic-based technologies. BMC Neurol. 2020 May 13;20(1):186. doi: 10.1186/s12883-020-01759-4. PMID 32404132